CLINICAL TRIAL: NCT05677217
Title: Clinical Feasibility of Nab-paclitaxel Plus Gemcitabine-cisplatin Chemotherapy in Patients With Locally Advanced Cholangiocarcinoma and Discovery of Biomarkers
Brief Title: Clinical Feasibility of Nab-paclitaxel Plus Gemcitabine-cisplatin Chemotherapy in Locally Advanced Cholangiocarcinoma
Status: Recruiting | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-11-002
Record Dates: First submitted 2022-11-16; First posted 2023-01-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and, if available, tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nab-paclitaxel plus gemcitabine-cisplatin: gemcitabine, 800 mg/m2, cisplatin, 25 mg/m2, and nab-paclitaxel, 100 mg/m2, on days 1 and 8 of 21-day cycles

SUMMARY:
The objective of this observational study is to identify patients with locally advanced cholangiocarcinoma treated with nab-paclitaxel and gemcitabine-cisplatin chemotherapy.

In this clinical study, peripheral blood and tumor tissues will be analyzed at baseline and every 3 cycles after systemic drug treatment in patients with locally advanced cholangiocarcinoma, and correlation with treatment was analyzed. This is an exploratory study to discover biomarkers that are highly correlated with treatment response.

DETAILED DESCRIPTION:
Although surgical treatment is the only treatment for cholangiocarcinoma, most patients are diagnosed at a metastatic or locally advanced stage, and palliative chemotherapy is the main treatment method for this group of patients.

Recently, with the introduction of gemcitabine, cisplatin, and nab-paclitaxel combination chemotherapy for locally advanced cholangiocarcinoma, the treatment response rate is improving, and the number of cases of downgrade to an operable state is increasing.

However, there are no prospective studies confirming the rate of conversion surgery after gemcitabine, cisplatin, and Nab-paclitaxel combination therapy in locally advanced cholangiocarcinoma. As a result of long-term follow-up, more than 30% of patients relapsed, so it is urgent to develop predictive biomarkers before surgery.

There are reports that tumor DNA (ctDNA) accurately predicts recurrence after surgical treatment. Using blood samples that are relatively easy to collect compared to biopsies, it is possible to quantitatively measure tumor burden and to evaluate the effectiveness of systemic treatments such as chemotherapy. It is a very popular tool for measuring and predicting the success of surgical treatment in advanced solid cancer.

The purpose of this study was to determine the rate of conversion surgery after treatment with Gemcitabine, Cisplatin, and Nab-paclitaxel in patients with inoperable locally advanced cholangiocarcinoma through an observational study. In addition, the purpose of this study is to verify the performance of biomarkers in predicting recurrence and survival after ctDNA and RNA conversion surgery in a situation where there is no clinical strategy to select a group of patients who can try radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Those above the age of 19 who understand the purpose of the study and agree to participate in the collection of samples during the study.
* Patients with histologically or cytologically confirmed inoperable locally advanced cholangiocarcinoma (gallbladder cancer, extrahepatic biliary tract cancer, intrahepatic biliary tract cancer)
* Patients who underwent an NGS test with advanced cholangiocarcinoma tissues
* Patients planning to be treated with nab-paclitaxel plus gemcitabine-cisplatin combination therapy
* ECOG performance status 0 or 1

Exclusion Criteria:

* Systemic condition accompanied by instability of vital signs such as infection or organ failure
* Patients who have previously received palliative chemotherapy for cholangiocarcinoma
* Those with mental/neurological conditions or dementia who have difficulties understanding and completing the consent form
* Those who are assessed as not suitable for this study, at the discretion of the researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of advanced cholangiocarcinoma patients through a competitive registration process at CHA Bundang Hospital, Haeundae Paik Hospital, and Seoul National University Bundang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Conversion Surgery Rate | 6 months
  Proportion of patients who underwent conversion surgery

SECONDARY OUTCOMES:
OS | 2 years
  Overall survival is calculated as the time from initiation of treatment until death.
  The follow-up period is from initiation of treatment until the date of death or for 1 year after last patient enrollment, whichever is earlier.
ORR | 1 year
  Overall Response Rate follow-up will be conducted every 6 weeks. Lesion will be evaluated according to RECIST 1.1 (CR, complete disappearance or LN short axis diameter < 1.0cm; PR, ≥30% reduction; PD, ≥20% increase; SD, neither CR, PR nor PD).
  The follow-up period is from initiation of treatment until date of disease progression or death or for 1 year after last patient enrollment, whichever is earlier.
PFS | 2 years
  Progression Free Survival is calculated as the time from initiation of treatment until the date of disease progression or death without PD.
  The follow-up period is from initiation of treatment until the date of disease progression or death without PD or for 1 year after last patient enrollment, whichever is earlier.
  Each time ORR is measured at 2-month intervals, progression-free survival will be checked.

OTHER OUTCOMES:
Recurrence Rate | through study completion, an average of 1 year
  Rate of recurrence after conversion surgery
Change of ctDNA | From baseline to 1 year of treatment
  The concentration of circulating DNA(ctDNA) in blood samples from patients with cholangiocarcinoma.
Identification of potential Biomarkers of Conversion Surgery | From baseline to 1 year of treatment
  Analysis of the expression patterns of immune-related proteins in tissue/blood samples collected in this study to identify biomarkers related to conversion surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD,PhD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarnagin WR, Fong Y, DeMatteo RP, Gonen M, Burke EC, Bodniewicz BS J, Youssef BA M, Klimstra D, Blumgart LH. Staging, resectability, and outcome in 225 patients with hilar cholangiocarcinoma. Ann Surg. 2001 Oct;234(4):507-17; discussion 517-9. doi: 10.1097/00000658-200110000-00010. PMID 11573044
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Kim BJ, Hyung J, Yoo C, Kim KP, Park SJ, Lee SS, Park DH, Song TJ, Seo DW, Lee SK, Kim MH, Park JH, Cho H, Ryoo BY, Chang HM. Prognostic factors in patients with advanced biliary tract cancer treated with first-line gemcitabine plus cisplatin: retrospective analysis of 740 patients. Cancer Chemother Pharmacol. 2017 Jul;80(1):209-215. doi: 10.1007/s00280-017-3353-2. Epub 2017 Jun 8. PMID 28597043
- [Background] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Background] Tie J, Cohen JD, Lahouel K, Lo SN, Wang Y, Kosmider S, Wong R, Shapiro J, Lee M, Harris S, Khattak A, Burge M, Harris M, Lynam J, Nott L, Day F, Hayes T, McLachlan SA, Lee B, Ptak J, Silliman N, Dobbyn L, Popoli M, Hruban R, Lennon AM, Papadopoulos N, Kinzler KW, Vogelstein B, Tomasetti C, Gibbs P; DYNAMIC Investigators. Circulating Tumor DNA Analysis Guiding Adjuvant Therapy in Stage II Colon Cancer. N Engl J Med. 2022 Jun 16;386(24):2261-2272. doi: 10.1056/NEJMoa2200075. Epub 2022 Jun 4. PMID 35657320
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Cheon J, Lee CK, Sang YB, Choi HJ, Kim MH, Ji JH, Ko KH, Kwon CI, Kim DJ, Choi SH, Kim C, Kang B, Chon HJ. Real-world efficacy and safety of nab-paclitaxel plus gemcitabine-cisplatin in patients with advanced biliary tract cancers: a multicenter retrospective analysis. Ther Adv Med Oncol. 2021 Aug 7;13:17588359211035983. doi: 10.1177/17588359211035983. eCollection 2021. PMID 34394748